CLINICAL TRIAL: NCT05700487
Title: THE EFFECT OF PELVIC FLOOR EXERCISES ON URINARY INCONTINENCE AND QUALITY OF LIFE AFTER PROSTATECTOMY
Brief Title: EFFECT ON QUALITY OF LIFE AFTER PROSTATECTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Assosc.Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PROSTATK
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: PROSTATECTOMY; URINARY INCONTINENCE
Keywords: Radical Prostatectomy; Pelvic Floor Exercises; Urinary Incontinence; Quality of life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The person applying the data sheets is an unbiased surveyor who does not know about the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in this group continued their routine medicaltreatmentprogram without any treatment
- Intervention Group (Experimental): Pelvic floor exercises (PTE) training in the preoperative period, regular PTE was performed three times a day for 6 months in the postoperative period, and the continuity of the exercises was checked by telephone
  Interventions: Other: PELVIC FLOOR EXERCISES

INTERVENTIONS:
Other: PELVIC FLOOR EXERCISES — Regular Pelvic floor exercises was performed three times a day for six months in the postoperative period
  Other Names: Intervention Group
  Arms: Intervention Group

SUMMARY:
Aim: This study was conducted to determine the effect of pelvic floor exercises (PTE) on urinary incontinence and quality of life (QOL) after radical prostatectomy (RP).

Methods: This randomized controlled, single-blind, experimental study was completed with a total of 33 RP patients, 18 of whom were interventions, and 15 were controls. The intervention group was given pelvic floor exercises (PTE) training in the preoperative period, regular PTE was performed three times a day for six months in the postoperative period, and the continuity of the exercises was checked by telephone. On the other hand, no intervention was applied to the control group other than routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Having the mental competence to understand the questions,
* Radical prostatectomy was performed due to the diagnosis of localized prostate cancer,
* Continuing post-operative follow-up,
* No incontinence problem before surgery,
* Anatomically free of genito-urinary system pathology,
* Those who volunteered to participate in the study were recruited.

Exclusion Criteria:

- With bladder insufficiency (dysfunction),

• Individuals with a different type of incontinence problem such as stress incontinence, neurogenic bladder were not included in the study.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients were included because it was after prostatectomy.
Enrollment: 33 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Quality of life Scale(SF-36) | The first measurement was made when the patients were included in the study.
  It measures the quality of life of individuals in 7 dimensions. These dimensions are physical function, social function, role limitations due to physical functions, role limitations due to emotional problems, mental health energy/vitality, pain and general perception of health. Instead of giving only a single total score, the scale is for each subscale. gives a total score separately. Subscales evaluate health from 0 to 100. "0 points" denotes the worst health condition, and "100 points" denotes the best health condition.
Quality of life Scale(SF-36) | It was performed at the 1st month follow-ups of the patients.
  It measures the quality of life of individuals in 7 dimensions. These dimensions are physical function, social function, role limitations due to physical functions, role limitations due to emotional problems, mental health energy/vitality, pain and general perception of health. Instead of giving only a single total score, the scale is for each subscale. gives a total score separately. Subscales evaluate health from 0 to 100. "0 points" denotes the worst health condition, and "100 points" denotes the best health condition.
Quality of life Scale(SF-36) | It was performed at the 3st month follow-ups of the patients.
  It measures the quality of life of individuals in 7 dimensions. These dimensions are physical function, social function, role limitations due to physical functions, role limitations due to emotional problems, mental health energy/vitality, pain and general perception of health. Instead of giving only a single total score, the scale is for each subscale. gives a total score separately. Subscales evaluate health from 0 to 100. "0 points" denotes the worst health condition, and "100 points" denotes the best health condition.
Quality of life Scale(SF-36) | It was performed at the 6st month follow-ups of the patients.
  It measures the quality of life of individuals in 7 dimensions. These dimensions are physical function, social function, role limitations due to physical functions, role limitations due to emotional problems, mental health energy/vitality, pain and general perception of health. Instead of giving only a single total score, the scale is for each subscale. gives a total score separately. Subscales evaluate health from 0 to 100. "0 points" denotes the worst health condition, and "100 points" denotes the best health condition.

SECONDARY OUTCOMES:
The Overactive Bladder (OAB-V8 ) | The first measurement was made when the patients were included in the study.
  Used to determine clinical incontinence. The OAB- V8 inquiry form determined the severity of the patients' complaints, none (0); very few (1); a little (2); quite a few (3); many (4); and it consists of 8 questions that can be graded as too many (5). The total score ranges from 0 to 40.
The Overactive Bladder (OAB-V8 ) | It was performed at the 1st month follow-ups of the patients.
  Used to determine clinical incontinence. The OAB- V8 inquiry form determined the severity of the patients' complaints, none (0); very few (1); a little (2); quite a few (3); many (4); and it consists of 8 questions that can be graded as too many (5). The total score ranges from 0 to 40.
The Overactive Bladder (OAB-V8 ) | It was performed at the 3st month follow-ups of the patients.
  Used to determine clinical incontinence. The OAB- V8 inquiry form determined the severity of the patients' complaints, none (0); very few (1); a little (2); quite a few (3); many (4); and it consists of 8 questions that can be graded as too many (5). The total score ranges from 0 to 40.
The Overactive Bladder (OAB-V8 ) | It was performed at the 6st month follow-ups of the patients.
  Used to determine clinical incontinence. The OAB- V8 inquiry form determined the severity of the patients' complaints, none (0); very few (1); a little (2); quite a few (3); many (4); and it consists of 8 questions that can be graded as too many (5). The total score ranges from 0 to 40.

OTHER OUTCOMES:
The Marmara Post-Prostatectomy Incontinence Symptom Score Form | The first measurement was made when the patients were included in the study.
  It determines how incontinence affects an individual's life. The survey consists of 8 questions and 3 parts. Point values between 0 and 28 can be obtained from the questionnaire. A high total score indicates an increase in the negative impact of incontinence on the patient.
The Marmara Post-Prostatectomy Incontinence Symptom Score Form | It was performed at the 1st month follow-ups of the patients.
  It determines how incontinence affects an individual's life. The survey consists of 8 questions and 3 parts. Point values between 0 and 28 can be obtained from the questionnaire. A high total score indicates an increase in the negative impact of incontinence on the patient.
The Marmara Post-Prostatectomy Incontinence Symptom Score Form | It was performed at the 3st month follow-ups of the patients.
  It determines how incontinence affects an individual's life. The survey consists of 8 questions and 3 parts. Point values between 0 and 28 can be obtained from the questionnaire. A high total score indicates an increase in the negative impact of incontinence on the patient.
The Marmara Post-Prostatectomy Incontinence Symptom Score Form | It was performed at the 6st month follow-ups of the patients.
  It determines how incontinence affects an individual's life. The survey consists of 8 questions and 3 parts. Point values between 0 and 28 can be obtained from the questionnaire. A high total score indicates an increase in the negative impact of incontinence on the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- ERciyes University, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Gacci M, Carini M, Simonato A, Imbimbo C, Gontero P, Briganti A, De Cobelli O, Fulcoli V, Martorana G, Nicita G, Mirone V, Carmignani G. Factors predicting continence recovery 1 month after radical prostatectomy: results of a multicenter survey. Int J Urol. 2011 Oct;18(10):700-8. doi: 10.1111/j.1442-2042.2011.02826.x. Epub 2011 Aug 11. PMID 21834853
- [Background] Almallah YZ, Grimsley SJ. A report of a regional service for post-prostatectomy urinary incontinence: a model for best practice? Ther Adv Urol. 2015 Apr;7(2):69-75. doi: 10.1177/1756287214561625. PMID 25829950
- [Background] Venderbos LDF, Aluwini S, Roobol MJ, Bokhorst LP, Oomens EHGM, Bangma CH, Korfage IJ. Long-term follow-up after active surveillance or curative treatment: quality-of-life outcomes of men with low-risk prostate cancer. Qual Life Res. 2017 Jun;26(6):1635-1645. doi: 10.1007/s11136-017-1507-7. Epub 2017 Feb 6. PMID 28168601
- [Background] Santa Mina D, Matthew AG, Hilton WJ, Au D, Awasthi R, Alibhai SM, Clarke H, Ritvo P, Trachtenberg J, Fleshner NE, Finelli A, Wijeysundera D, Aprikian A, Tanguay S, Carli F. Prehabilitation for men undergoing radical prostatectomy: a multi-centre, pilot randomized controlled trial. BMC Surg. 2014 Nov 13;14:89. doi: 10.1186/1471-2482-14-89. PMID 25394949
- [Background] Lee EW, Kobashi KC. Mixed incontinence: what takes precedence in its management? Curr Urol Rep. 2014 Dec;15(12):461. doi: 10.1007/s11934-014-0461-y. PMID 25287258